CLINICAL TRIAL: NCT04842812
Title: Engineered TILs/CAR-TILs With PD1 Knockout and Anti-PD1/CTLA4-scFv Secreting or CARs Against Various Antigens to Treat Advanced Solid Tumors
Brief Title: Engineered TILs/CAR-TILs to Treat Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Guangdong Zhaotai InVivo Biomedicine Co. Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZZTIL-012
Record Dates: First submitted 2021-04-04; First posted 2021-04-13 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Liver Cancer; Lung Cancer; Breast Cancer; Colo-rectal Cancer; Brain Tumor; Solid Tumor, Adult; PD1; CTLA4
Keywords: liver Cancer; Lung Cancer; Solid Tumor; TIL; CAR-TIL; PD1; CTLA4; GPC3; Mesothelin; B7-H3; CRISPRA-CAS9
MeSH Terms: conditions — Liver Neoplasms; Lung Neoplasms; Breast Neoplasms; Colonic Neoplasms; Brain Neoplasms | interventions — Mesothelin; PSCA protein, human

STUDY DESIGN:
Intervention Model Description: TILs treatment of solid cancers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TILs/CAR-TILs treatment (Experimental): Obtain TILs/CAR-TILs from advanced solid tumor patients and infuse them back to evaluate safety and clinical efficacy of the treatment.
  Interventions: Biological: TILs and CAR-TILs targeting HER2, Mesothelin, PSCA, MUC1, Lewis-Y, GPC3, AXL, EGFR, Claudin18.2/6, ROR1, GD1, or B7-H3

INTERVENTIONS:
Biological: TILs and CAR-TILs targeting HER2, Mesothelin, PSCA, MUC1, Lewis-Y, GPC3, AXL, EGFR, Claudin18.2/6, ROR1, GD1, or B7-H3 — TILs and CAR-TILs injection: 1-10×10e7/kg cells for each treatment; 3 or more cycles.

SUMMARY:
Tumor infiltration lymphocytes (TILs) have been harvested from advanced cancer patients and constructed to knockout PD1 gene and express scFvs against both PD1 and CTALA4 and CARs against various antigens, followed by transfusion into the patients. The safety, tolerance, and preliminary clinical efficacy of the TILs will be evaluated.

DETAILED DESCRIPTION:
1. Choose appropriate patients with advanced lung or other cancers, with written consent for this study;
2. Perform biopsy or collect cancerous effusion in thorax or abdomen to obtain TILs by standard protocol;
3. Grow TILs and engineered the tumor-effective TILs with CRISPRA-CAS9 technique to knockdown PD1 and electronic-transfection strategy to express scFvs that target PD1 and CTLA4; amplify the engineered T cells as needed, test the quality and killing activity of the TILs and then transfuse them back the patients via systemic or local injections via standard protocol, and follow up closely to collect related parameters as needed;
4. To enhance the killing capability, tumor-noneffective TILs have also been genetically engineered to express various CARs targeting HER2/Mesothelin/Lewis-Y/PSCA/MUC1/ GPC3/AXL/EGFR/Claudin18.2/B7-H3/ROR1/GD2/AXL/Claudin6-DAP10 with knockdown of PD1/HPK1 as appropriate;
5. Evaluate the clinical results as needed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced cancers that failed to current available therapies;
2. Life expectancy >12 weeks;
3. Adequate heart, lung, liver, kidney functions;
4. Available for tumor biopsy or cancerous effusions;
5. Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent.

Exclusion Criteria:

1. Had accepted gene therapy before;
2. Severe virus infection such as HBV, HCV, HIV, et al; Known HIV positivity;
3. Active infectious disease related to bacteria, virus, fungi, et al;
4. Other severe diseases that the investigators consider not appropriate;
5. Pregnant or lactating women;
6. Systemic steroid treatment (greater than or equal to 0.5 mg prednisone equivalent/kg/day);
7. Other conditions that the investigators consider not appropriate.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Safety of TILs/CAR-TILs treatment in advanced solid cancers | up to 36 months
  Assessing Number of participants with treatment-related adverse events as assessed by CTCAE v4.0.

SECONDARY OUTCOMES:
Primary clinical efficacy of the TILs/CAR-TILs treatment in advanced solid cancers | 15 years
  Assessing various clinical response rates including complete response, partial response, stable disease, and progress disease during and after TILs/CAR-TILs treatment in advanced solid cancers.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenfeng Zhang, MD, PhD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No